CLINICAL TRIAL: NCT07204288
Title: LUMBAR & SACROILIAC FUSION STUDY: MULTI-CENTER PROSPECTIVE RADIOGRAPHIC STUDY ON SUBJECTS PREVIOUSLY IMPLANTED WITH SPINAL SIMPLICITY LUMBAR AND/OR SACROILIAC FUSION DEVICE(S)
Brief Title: LUMBAR & SACROILIAC FUSION STUDY
Acronym: FUSION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Simplicity LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SSMMSI-2025-CIP
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fusion of Spine; Sacroiliac; Fusion

STUDY DESIGN:
Intervention Model Description: This will involve patients previously commercially implanted with Minuteman G5 MIS fusion plate, the Liberty sacroiliac fusion device, and/or the Patriot sacroiliac fusion device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Previously implanted with lumbar and/or sacroiliac fusion device(s) (Other): This study will involve patients previously commercially implanted with Minuteman G5 MIS fusion plate, the Liberty sacroiliac fusion device, and/or the Patriot sacroiliac fusion device. Subjects will undergo a CT scan, if applicable and PROs.
  Interventions: Other: Cat Scan, if applicable

INTERVENTIONS:
Other: Cat Scan, if applicable — Cat Scan is being used to assess fusion in previously implanted population

SUMMARY:
This study is a multi-center, observational, prospective and retrospective data collection study

DETAILED DESCRIPTION:
The purpose of this study is to evaluate fusion outcomes and patient-reported outcomes for Spinal Simplicity's lumbar and/or sacroiliac fusion implants: the Minuteman G5 MIS fusion plate, the Liberty sacroiliac fusion device, and/or the Patriot sacroiliac fusion device. This will involve identifying patients previously implanted with any of these devices and conducting both retrospective and prospective data collection/analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older at the time of enrollment
2. Be willing and able to provide informed consent and comply with study visit requirements
3. Subjects who received a Spinal Simplicity fusion implant(s) (Minuteman G5, Liberty, and/or Patriot) between April 1, 2022 and March 31, 2025

Exclusion Criteria:

1. Unable to provide consent and complete prospective data collection
2. Women who are pregnant, or may become pregnant, during the course of the study
3. Contraindication to CT scanning, in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Investigate radiographic outcomes | Enrollment
  The primary endpoints include the rate of fusion, and the rate of complications or reoperations.
  Fusion Scale:1) Radiographically evaluate the rate of fusion, as determined by a panel of independent radiologists per the below fusion assessment metrics: Lumbar fusion grading scale (Minuteman G5): 1- Definitely fused 2- Probably fused 3- Probably not fused 4- Definitely not fused;
  Sacroiliac fusion assessment (Liberty, Patriot):
  Device(s) will be evaluated for (i) the presence of bridging bone from ilium to sacrum; and (ii) any evidence of migration or loosening
  Additionally, if Minuteman G5 subjects have an interbody fusion device, interbody fusion will be assessed using the Bridwell scale:
  1- Definite fusion 2- Probable fusion 3- Intermediate fusion/possible motion 4- Pseudoarthrosis/no bony connection

SECONDARY OUTCOMES:
NRS/ Numeric Rating Scale | Enrollment
  1. Pain (Overall, Back and Leg) using NRS/numeric rating scale Overall pain, as well as back pain when standing/walking and leg pain when standing will be assessed using a numeric rating scale (NRS). The NRS is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
ODI/ Oswestry Disability Index | Enrollment
  Oswestry Disability Index (ODI) ODI is a self-reported questionnaire widely used to track changes in a patient's condition over time and evaluate the effectiveness of treatments for low back pain. The ODI consists of 10 sections, each addressing a specific aspect of daily functioning. A higher score indicates greater disability. The final score/index ranges from 0-100 scale. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed bound.
PGIC/ Patient Global Impression of Change | Enrollment
  The Patient Global Impression of Change (PGIC) PGIC is a standardized tool designed to assess a patient's self-reported perception of improvement or worsening in their health status over time. The PGIC consists of 1 question, using a 1 to 7 scale: 1-Very Much Improved to 7-Very much Worse.
Subject Satisfaction Survey | Enrollment
  Subject Satisfaction Survey Subject Satisfaction Survey is made up of 8 questions designed to assess a patient's self-reported satisfaction or dissatisfaction on a Likert scale. The Likert scale consists of 8 questions individually scored on a 1 to 5 scale: With lower scores indicating higher satisfaction and higher scores indicating greater dissatisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hedman, PhD, Study Chair — Spinal Simplicity LLC
Locations (3):
- United States (3):
  - Crimson Pain Management, Overland Park, Kansas
  - Nuroscience Research Center, Overland Park, Kansas
  - Nura Precision Pain Management, Edina, Minnesota

IPD SHARING:
Plan to Share IPD: No
Results will be published at the sponsor's discretion.